CLINICAL TRIAL: NCT04890405
Title: Clinical Comparative Study of Precision Flora Transplantation and Standardized Fecal Microbiota Transplantation in Patients With Irritable Bowel Syndrome.
Brief Title: Clinical Study of Selective Fecal Microbiota Transplantation in the Treatment of Irritable Bowel Syndrome.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yanling Wei (Other)
Responsible Party: Sponsor-Investigator, Yanling Wei, Department of Gastroenterology, Da ping Hospital, The Third Military Medical University, Third Military Medical University
Organization: Third Military Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TMMU-DP-GI-JZ-001
Record Dates: First submitted 2021-05-05; First posted 2021-05-18 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Irritable Bowel Syndrome Variant of Childhood
Keywords: irritable bowel syndrome; diarrhea; Fecal Microbiota Transplantation
MeSH Terms: conditions — Irritable Bowel Syndrome; Diarrhea

STUDY DESIGN:
Intervention Model Description: Diarrhea-type irritable bowel syndrome patients were randomly divided into 2 groups, and each group was given a different treatment method
Who Masked: Outcomes Assessor
Masking Description: The assessor of the scale does not know the grouping of patients when assessing the patient.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FMT group (Active Comparator): Standardized FMT once.Extract all the flora from the feces provided by the donor to make fecal bacteria transplant capsules. The patient took orally on an empty stomach, each time using 3.2g of fecal bacteria.
  Interventions: Procedure: Standardized FMT
- JZ group (Experimental): 1.6g Po perday,for 28 days. probiotics that are effective against diarrhea were selected to make precise flora capsules, which are taken when the patient is on an empty stomach, once a day, using 1.6 g of bacteria per day, orally for 28 consecutive days.
  Interventions: Combination Product: Precision Flora Transplantation

INTERVENTIONS:
Procedure: Standardized FMT — The group includes 35 patients. They will receive standardized FMT. Fecal bacteria capsules are used for fecal bacteria transplantation, 16 capsules are used each time, each capsule contains 200mg of fecal bacteria, and it is used orally. It was given only once.
  Arms: FMT group
Combination Product: Precision Flora Transplantation — The group includes 35 patients. They will receive Precision Flora Transplantation. They were used self-developed precision transplant capsules for precision flora transplantation. 4 capsules are used each time. Each capsule contains 400mg of various probiotics effective against diarrhea. It is used orally, once a day,for 28 days.
  Arms: JZ group

SUMMARY:
In order to seek a more precise and convenient treatment, we made a self-made precise transplant capsule that is effective against diarrhea. Compared with standardized fecal microbiota transplantation transplantation on the treat of diarrhea-type irritable bowel syndrome. To observe the similarities and differences of the effect between the two treatment methods on the disease. and the changes in intestinal bacteria was also observed.

DETAILED DESCRIPTION:
In order to clarify the effectiveness of precision fecal bacteria transplantation, we have independently developed precision transplantation capsules. Seventy patients with diarrhea-type irritable bowel syndrome were selected and randomly divided into 2 groups. The patients in the first group were treated with standard fecal bacteria transplantation once, and the patients in other group were treated with precision transplantation capsules for 28 days. The clinical symptoms of the patients of the two groups were observed before and 2, 4, 8, 12, 24, and 48 weeks after the treatment, and stool samples were collected for intestinal flora detection. The purpose is to observe and compare the efficacy of the two treatment methods and their influence on the intestinal flora.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18 ~ 75 years.
* Patients who meet the diagnostic criteria of Rome IV of Irritable Bowel Syndrome and are definitely diagnosed as IBS-D.
* IBS has been diagnosed for more than 6 months, and has been treated with conventional drugs without obvious curative effect or repeated attacks.
* No other serious diseases, no mental disorders, and normal communication skills.
* Sign informed consent and agree to participate in this study.
* No antibiotics and probiotics were used within one month.

Exclusion Criteria:

* Patients are unwilling to participate in this study.
* Other serious diseases of heart, liver, kidney, respiration, digestion, blood and endocrine system.
* Combined with intestinal double infection, such as CDI, enterohemorrhagic Escherichia coli, Salmonella, Shigella, Campylobacter, plague, cytomegalovirus, etc.
* Liver function is significantly abnormal or has the following history of liver disease: AST or ALT is higher than 2 times of the upper limit of normal value, history of liver cirrhosis and hepatic encephalopathy, history of esophageal varices or history of portal shunt.
* There is evidence of renal function damage or the following history of kidney disease: serum creatinine is 1.5 times higher than the upper limit of normal value; History of dialysis; Or a history of nephrotic syndrome.
* Patients with various acute infections, tumors, severe arrhythmia, mental system disorders, and drug or alcohol addicts.
* History of abdominal surgery (except appendicitis, cholecystitis, caesarean section and hysterectomy).
* Those who were allergic to capsule drugs or contraindications.
* Lactose intolerance.
* Clinical researchers who are engaged in other related irritable bowel syndrome at the time of enrollment or within 3 months before enrollment.
* It is difficult to complete the follow-up, or various factors affecting the compliance.
* Pregnant or lactating women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-05-20 (Estimated); Primary Completion 2021-10-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
IBS-SSS score | 12 Week after treatment
  Severity of irritable bowel syndrome.The score varies from 0 to 500. Higher scores suggest more severe condition.

SECONDARY OUTCOMES:
Clinical remission rate | 2、4、8、12 Week after treatment
  Proportion of people in clinical remission after treatment
GSRS score | 0、2、4、8、12Week after treatment
  Gastrointestinal Symptom Rating Scale.The score varies from 16 to 112. Higher scores suggest more severe gastrointestinal pathology.
IBS-QoL score | 0、2、4、8、12Week after treatment
  Quality of life score for IBS patients.The score varies from 0 to 136. Higher scores suggest greater impact of disease on life
PHQ-9 | 0、2、4、8、12Week after treatment
  Patient Health Questionnaire-9.The score varies from 0 to 27. Higher scores suggest more severe the depression
GAD-7 | 0、2、4、8、12Week after treatment
  Generalized Anxiety Scale-7.The score varies from 0 to 21. Higher scores suggest heavier the anxiety.
SAS | 0、2、4、8、12Week after treatment
  Self-rating Anxiety Scale.The score varies from 25 to 100. Higher scores suggest greater degree of anxiety.
SDS | 0、2、4、8、12after treatment
  Self-rating Depression Scale.The score varies from 25 to 100. Higher scores suggest more severe depression.
Intestinal flora | 0、2、4、8、12Week after treatment
  Use metagenomics technology to detect intestinal flora

CONTACTS AND LOCATIONS:
Overall Officials: Yanling Wei, Principal Investigator — Army Medical Center of PLA